CLINICAL TRIAL: NCT02807493
Title: Use of an Occlusal Support Device During the Second Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DENT-2016-23918
Record Dates: First submitted 2016-06-08; First posted 2016-06-21 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Pregnancy
Keywords: Pregnancy; Labor and Delivery; Occlusal Support Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Occlusal Support Device (Experimental): Support device for women in labor
  Interventions: Device: Occlusal Support Device
- Control (Placebo Comparator): No device given for women in labor
  Interventions: Other: Control

INTERVENTIONS:
Device: Occlusal Support Device — Bite plate
  Arms: Occlusal Support Device
Other: Control — Control group
  Arms: Control

SUMMARY:
The primary objectives of this study are to determine if the use of an Occlusal Support Device (OSD)(Mouthguard) can reduce the duration and intensity of the second stage of labor, reduce the incidence of labor complications including Caesarian Sections and improve Apgar scores in newborns

DETAILED DESCRIPTION:
Prolonged labor, especially during the second stage of active expulsive effort (the pushing phase), is associated with increased risk of maternal complications (e.g. tissue trauma, postpartum hemorrhage, intra-amniotic infection). Developing an effective method to assist and maximize maternal expulsion effort should be of great value in reducing the number of complications, also including cesarean section or instrumental deliveries. Past studies published in the dental literature have shown that specially designed oral appliances that support the dental occlusion may increase the isometric strength of different muscle groups. Increased strength of the neck muscles could improve efficiency of the Valsalva maneuver in increasing intra-uterine pressure, and thus decreasing the duration of phase II of labor. Nulliparous women with uncomplicated singleton pregnancy will be randomly assigned to either the study group (Dental appliance) or the no dental appliance group. Duration of labor will be measured for both phase I and phase II. Rates for cesarean section and instrument deliveries and other complications will be charted as well as Apgar scores .

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Uncomplicated pregnancy
* Singleton pregnancy

Exclusion Criteria:

* Unable to provide informed consent or comply with study protocol,
* High risk and/or complicated pregnancy,
* Have multiple fetuses as diagnosed by ultrasound,
* Have extensive decay or multiple broken/missing teeth that will interfere with the fabrication of an OSD

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 347 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Gambucci, DDS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Occlusal Support Device | Control
Started | 174 | 173
Completed | 87 | 121
Not Completed | 87 | 52
Not completed — Adverse Event | 5 | 2
Not completed — Lost to Follow-up | 6 | 0
Not completed — Physician Decision | 4 | 1
Not completed — Protocol Violation | 7 | 0
Not completed — Withdrawal by Subject | 17 | 10
Not completed — Other withdrawal | 17 | 0
Not completed — C-Section Prior to Stage 2 of Labor | 31 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Occlusal Support Device | Control | Total
Number analyzed (Participants) | 174 | 173 | 347
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 174 | 173 | 347
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 173 | 347
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 17 | 19 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 11 | 22
  White | 134 | 126 | 260
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 9 | 16 | 25

OUTCOME MEASURES:

1. Primary Outcome: Stage 2 Duration of Labor
Description: Determine if an Occlusal Support Device (OSD) can reduce the duration of the second stage of labor
Time Frame: Duration of labor
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Occlusal Support Device | Control
Number analyzed (Participants) | 75 | 106
minutes | 120.2 (88.2) | 107 (83.9)

2. Primary Outcome: Number of Participants With a Cesarian Section
Description: Determine if an OSD can reduce the incidence of labor complications including Caesarian Sections
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Occlusal Support Device | Control
Number analyzed (Participants) | 87 | 121
participants | 12 | 13

3. Primary Outcome: Average Apgar Score
Description: Determine if the use of an OSD can improve Apgar scores in newborns. The Apgar test is done by a doctor, midwife, or nurse. The provider examines the baby's:
  Breathing effort Heart rate Muscle tone Reflexes Skin color Each category is scored with 0, 1, or 2, depending on the observed condition. Higher scores are better. Scores are added for a total ranging from 0-10.
Time Frame: at minute 1 and minute 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Occlusal Support Device | Control
Number analyzed (Participants) | 87 | 121
score on a scale
  APGAR at min 1 | 7.8 (1.6) | 7.9 (1.4)
  APGAR at min 5 | 8.8 (0.5) | 8.8 (0.7)

ADVERSE EVENTS:
Time Frame: Duration of labor
Arm/Group | Occlusal Support Device | Control
All-Cause Mortality (participants affected / at risk) | 0/174 | 0/173
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/173
Other Adverse Events (participants affected / at risk) | 5/174 | 2/173
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Occlusal Support Device (N=174) | Control (N=173)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT02807493/Prot_SAP_006.pdf
  • Informed Consent Form (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT02807493/ICF_003.pdf